CLINICAL TRIAL: NCT02391129
Title: Locking Compression Plate Fixation Versus Revision- Prosthesis of Vancouver-B2, B3 and C Periprosthetic Femoral Fractures After Total Hip Replacement
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Julian Joestl, MD, Medical University of Vienna
Other Study IDs: 1674/2014
Record Dates: First submitted 2015-03-07; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Periprosthetic Fractures
MeSH Terms: conditions — Periprosthetic Fractures | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Hyperion Prosthesis: Patients treated with the second generation long-stem revision prosthesis
  Interventions: Procedure: Operation for Periprosthetic fractures of the hip with stem loosening
- Helios Prosthesis: Patients treated with the first generation long-stem revision prosthesis
  Interventions: Procedure: Operation for Periprosthetic fractures of the hip with stem loosening
- Locking compression plate: Patients treated with LCP
  Interventions: Procedure: Operation for Periprosthetic fractures of the hip with stem loosening

INTERVENTIONS:
Procedure: Operation for Periprosthetic fractures of the hip with stem loosening

SUMMARY:
The purpose of this study was to compare the clinical (range of motion, weight bearing, quality of life) and radiographic outcome (boney consolidation) between open reduction and internal fixation using locking compression plates with revision prosthesis using a non-cemented long femoral stem in a group of patients with a Vancouver type-B2, B3 and C periprosthetic fracture after primary total hip replacement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Vancouver type- BlI, BIII and C fractures and unstable femoral prosthesis stem.

Exclusion Criteria:

* Patients with pathological fractures,
* Vancouver type-A, Bl, and
* stable femoral prosthesis stem,
* Patients with hemi - prosthesis and periprosthetic femoral fractures were excluded from final analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We retrospectively reviewed a consecutive series of 102 patients with Vancouver type-B2, B3 and C periprosthetic fractures and unstable femoral stem, which had been prospectively entered, in our hip-trauma database.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome (Range of Motion of the hip) | follow up of at least 1 year
  Range of Motion of the hip
Radiographic Outcome (boney consolidation of the fracture) | follow up of at least 1 year
  boney consolidation of the fracture after 3 month, 6 month and at least 1 year after the operation

SECONDARY OUTCOMES:
Patient's Mobility (assessed by the Parker's Mobility Score) | follow up of at least 1 year
  Patient's Mobility assessed by the Parker's Mobility Score